CLINICAL TRIAL: NCT05690360
Title: Evaluation of the Pregnancy Outcomes and Time to Embryo Transfer Regarding the Progesterone Levels of Natural Cycle-FETs
Brief Title: Pregnancy Outcomes of Patients Having NC-FET Regarding the Progesterone Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nazli Albayrak, Resident in training at Acibadem University, School of Medicine, Department of Obstetrics and Gynecology, Acibadem University
Other Study IDs: 2022-17/60
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We recently identify in our previous study 'NCT052115832' the progesterone levels for the embryo transfer in natural thaw cycles. Since it is shown that progesterone levels work better than LH levels in order to detect the time to transfer, we aimed to show the pregnancy outcomes of the natural thaw cycles which had the transfer date regarding the progesterone levels.

ELIGIBILITY:
Inclusion Criteria:

* patients with regular menstrual cycle
* patients aged btw 20-40
* patients with pregnancy with NC-FET by using the progesterone for the detection of ovulation

Exclusion Criteria:

* Spontenous pregnancies
* Multiple pregnancies

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Participants are going to be selected from the patients who applied to infertility clinic, and are pregnant with in vitro fertilization natural cycle- frozen embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Cummulative Live Birth Rate | 10 months
  Live birth rates of Patient with NC-FET followed up with progesterone levels
Biochemical pregnancy results | 2 months
  Biochemical pregnancy results of patients with NC-FET followed up with progesterone levels
Pregnancy complications | 10 months
  Obstetric Complications of Patient with NC-FET followed up with progesterone levels

CONTACTS AND LOCATIONS:
Overall Officials: NAZLI ALBAYRAK, MD, Principal Investigator — Acıbadem University School of Medicine; TURGUT AYDIN, MD, Principal Investigator — Acıbadem University School of Medicine; NADIYE KOROGLU, MD, Principal Investigator — Acıbadem University School of Medicine
Locations (1):
- Acibadem University Atakent Hospital, Istanbul, Turkey (Türkiye)